CLINICAL TRIAL: NCT00764829
Title: Blood Samples to Evaluate Biomarkers of Donor Chimerism
Status: Completed | Type: Observational
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Jeannine S. McCune, PharmD, Fred Hutchinson Cancer Research Center
Other Study IDs: FHCRC - 1980.00; R01HL091744 (NIH); IR-5957 (Other: FHCRC)
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Leukemia; Hodgkins Disease; Non-hodgkins Lymphoma; Myelodysplastic Syndrome
Keywords: hematopoietic stem cell transplantation; fludarabine; mycophenolate mofetil; mycophenolic acid; biomarkers
MeSH Terms: conditions — Leukemia; Hodgkin Disease; Lymphoma, Non-Hodgkin; Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma,DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
We are interested in patient-specific factors that may affect the balance of recipient cells and donor cells in patients who receive stem cell transplants. We will look at the way the patient's body breaks down two drugs, fludarabine and mycophenolate mofetil, and how these two drugs affect the patient's body.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a hematologic disease or malignancy
* Scheduled to receive nonablative conditioning with fludarabine and total body irradiation
* Donor is well-matched by high resolution DNA techniques.
* Scheduled to receive postgrafting immunosuppression of oral MMF (CellCept) and an oral calcineurin inhibitor.
* Age >18 years at the time of enrollment.

Exclusion criteria:

-Diagnosed with an immunodeficiency disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hematopoietic stem cell transplant patients receiving fludarabine and mycophenolate mofetil.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2008-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Donor T-cell chimerism | Day 28 post-transplant

SECONDARY OUTCOMES:
Exposure to fludarabine and mycophenolate mofetil and their breakdown products. | Before and after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Jeannine S McCune, PharmD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States